CLINICAL TRIAL: NCT01458145
Title: Minding the Baby Home Visiting: Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17098; R01HD057947 (NIH)
Record Dates: First submitted 2011-10-03; First posted 2011-10-24 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Attachment; Child Maltreatment; Maternal Sensitivity; Infant Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Home visits (Experimental)
  Interventions: Behavioral: Minding the Baby Home Visiting Program
- routine primary care at community health center (No Intervention)

INTERVENTIONS:
Behavioral: Minding the Baby Home Visiting Program — Weekly home visits for one year followed by bi-weekly home visits until child is 24 months of age provided to young at risk families by a team of nurse practitioner and social worker home visitors
  Arms: Home visits

SUMMARY:
This is an efficacy study of an intensive home visitation intervention, "Minding the Baby" (MTB). This reflective parenting program (aimed at enhancing maternal reflective capacities), is focused on first-time young mothers and infants living in an urban community. The study, grounded in attachment and human ecology theories integrates advanced practice nursing and mental health care by pairing master's level nurse practitioners and social workers with at-risk young families. Aims of the study are: 1) to determine the efficacy of the MTB intervention in young mothers and infants with respect to a) maternal outcome variables including the quality of the mother-infant relationship, maternal reflective capacities, maternal mastery/self-efficacy, parental competence, and maternal health and life course outcomes (educational success, employment, delaying subsequent child-bearing); and b) infant outcome variables including early attachment, infant health, and developmental outcomes; 2) to monitor fidelity and dose of the program with young mothers; 3) to describe the evolution of reflective capacities in adolescent mothers (contrasting intervention group with control group) through descriptive qualitative analyses of transcribed Pregnancy Interviews and Parent Development Interviews at the last trimester of pregnancy and at 24 months; 4) to conduct cost-effectiveness analyses of the program. The longitudinal two-group study (subjects nested within randomly assigned groups), will include multi-method (self report, interview and direct observation and coding of behaviors) approaches with a cohort of first-time multi-ethnic mothers between the ages of 14-25 (and their infants). MTB home visits occur weekly for intervention families (n=69) beginning in mid pregnancy and continuing through the first year, and then bi-weekly through the second year. Mothers and infants (n=69) in the control group will receive standard prenatal, postpartum and pediatric primary care in one of two community health centers (as will the intervention group) and also receive monthly educational materials about child health and development mailed to their homes. Maternal and infant outcome variables will be followed over time (pregnancy, 4, 12, and 24 months) as well as compared between the 2 groups. Cost analyses and analysis of the dose and sample characteristics linked to efficacy, will allow us to plan for translation of the model into clinical care and community sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Having a first child
* Speak English
* Obtains primary care from community health centers

Exclusion Criteria:

* No psychoses or terminal illnesses

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maternal reflective capacities | 27 months
  Coded interview data from Pregnancy Interviews in third trimester and Parent Development Interviews at 24 months.
Infant Attachment | 14 months
  Attachment pattern of child as measured by Strange Situation Procedure
Maternal life course outcomes | 24 months
  Ability to delay rapid subsequent childbearing within 24 months of first child's birth
child abuse or neglect | 24 months
  Reports of an open case with child protective services for parents and children within the study; documented by interview and health record

SECONDARY OUTCOMES:
Dose of intervention | 24 months
  Frequency, duration and content of home visits during the intervention
cost analysis for the program | 27 months
  cost analysis of program and outcomes regarding health and health service use
Description of reflective functioning in pregnant adolescents | baseline
  qualitative analysis of Pregnancy Interview transcripts from adolescent participants in third trimester of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Lois S Sadler, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Fair Haven Community Health Center, New Haven, Connecticut
  - Cornell Scott Hill Health Center, New Haven, Connecticut

REFERENCES:
- [Background] Flaherty SC, Sadler LS. A review of attachment theory in the context of adolescent parenting. J Pediatr Health Care. 2011 Mar-Apr;25(2):114-21. doi: 10.1016/j.pedhc.2010.02.005. Epub 2010 May 1. PMID 21320683
- [Background] Sadler LS, Newlin KH, Johnson-Spruill I, Jenkins C. Beyond the medical model: interdisciplinary programs of community-engaged health research. Clin Transl Sci. 2011 Aug;4(4):285-97. doi: 10.1111/j.1752-8062.2011.00316.x. PMID 21884518
- [Derived] Londono Tobon A, Condon E, Slade A, Holland ML, Mayes LC, Sadler LS. Participation in an Attachment-Based Home Visiting Program Is Associated with Lower Child Salivary C-Reactive Protein Levels at Follow-Up. J Dev Behav Pediatr. 2023 May 1;44(4):e292-e299. doi: 10.1097/DBP.0000000000001180. PMID 37126599